CLINICAL TRIAL: NCT06227195
Title: Mechanism of IL-10 Pathway-mediated Regulatory B Cell Dysfunction in Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Shufeng Li (Other)
Responsible Party: Sponsor-Investigator, Shufeng Li, Chief Physician, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: 2018S0097
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our previous work has shown that Treg function is impaired in OA patients, but the cause of Treg deficiency has not been investigated. Since Breg has been shown to promote Treg differentiation and tissue repair, it is highly likely that the absence of the immunomodulatory effect of Breg in OA patients leads to impaired Treg differentiation. Based on the above data, we hypothesized that Breg plays a protective role in the course of OA by regulating T cell composition and promoting Treg differentiation through the secretion of anti-inflammatory factor IL-10

ELIGIBILITY:
Inclusion Criteria:Patients who met the American College of Rheumatology diagnostic criteria for OA

-

Exclusion Criteria:

* Patients with trauma, other forms of arthritis such as rheumatoid arthritis, psoriatic arthritis or spondyloarthritis, and other active inflammatory diseases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee osteoarthritis come to our hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Breg | 4 and 8 weeks after DMM
  Regulatory B cells

SECONDARY OUTCOMES:
Cytokine secretion by T cells | 4 and 8 weeks after DMM
  Regulatory T cells

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China